CLINICAL TRIAL: NCT07165418
Title: A Multicenter, Randomized Controlled Study Comparing Vorolanib Tablets Plus Everolimus With Sunitinib in Patients With Advanced Renal Cell Carcinoma Who Have Progressed on Immunotherapy Monotherapy or in Combination With TKI
Brief Title: A Comparison of Vorolanib Tablets Combined With Everolimus Versus Sunitinib in Patients With Advanced Renal Cell Carcinoma Who Have Progressed After Treatment With Immunotherapy Monotherapy or in Combination With TKI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun GUO, Associate Director of Peking University Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ61
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vorolanib Tablets+Everolimus (Experimental)
  Interventions: Drug: Vorolanib Tablets+Everolimus
- Sunitinib (Active Comparator)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Vorolanib Tablets+Everolimus — Subjects received oral vorinib 200 mg once daily (QD) plus everolimus 5 mg once daily (QD), administered within 30 minutes after breakfast daily. Treatment cycles lasted 28 days and continued until disease progression.
  Arms: Vorolanib Tablets+Everolimus
Drug: Sunitinib — Subjects received oral sunitinib 50 mg once daily (QD) in a 4-week on, 2-week off regimen or a 2-week on, 1-week off regimen until disease progression.
  Arms: Sunitinib

SUMMARY:
This study is a multicenter, open-label, randomized controlled trial that enrolled 116 patients with advanced or metastatic renal cell carcinoma who had failed first-line treatment with PD-1/PD-L1 monotherapy or VEGFR TKI combined with PD-1/PD-L1 therapy. Patients were randomly assigned in a 1:1 ratio to receive either the experimental group treatment with vorolanib tablets combined with everolimus or the control group treatment with sunitinib as second-line therapy until disease progression. The study aimed to evaluate the efficacy and safety of vorolanib tablets combined with everolimus as second-line therapy for renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed renal clear cell carcinoma (histological or cytological);
2. Subjects who have failed prior treatment with a single anti-PD-1/PD-L1 agent or a combination of anti-PD-1/PD-L1 and anti-VEGFR TKI;
3. Age 18 to 80 years;
4. Estimated survival exceeding 12 weeks;
5. KPS score ≥70;
6. At least one measurable lesion per RECIST 1.1 criteria, which has not received prior radiation therapy;
7. Adequate organ function levels;
8. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization; all enrolled subjects (male or female) must use effective barrier contraception throughout treatment and for 4 weeks post-treatment;
9. Subjects must be capable of understanding and voluntarily signing the informed consent form, which must be signed prior to any trial procedures.

Exclusion Criteria:

1. Patients who have received one or more prior systemic anticancer treatment regimens for clear cell renal cell carcinoma;
2. Patients who have not previously received immunosuppressive therapy for advanced renal cell carcinoma;
3. Subjects currently undergoing anticancer therapy (excluding local radiotherapy for bone metastases);
4. Subjects with known hypersensitivity to similar drugs;
5. Subjects with active infectious diseases;
6. Any uncontrolled clinical condition;
7. Undergone major surgery within 4 weeks prior to enrollment;
8. History of significant psychiatric disorders that may impair understanding of informed consent or compliance with the study protocol;
9. Any condition affecting the subject's ability to swallow medication;
10. Pregnant or lactating women;
11. Subjects with severe pulmonary disease, asthma, or COPD history, with pulmonary function tests indicating moderate or greater impairment;
12. Any other factors deemed by the investigator to make the subject unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | The time from study entry to the first disease progression (PD) or death .Estimate up to 2 years.
  The time from study entry to the first disease progression (PD) or death from any cause, as assessed by the investigator.

SECONDARY OUTCOMES:
Overall Survival（OS） | The duration of treatment is determined from the start date to the date of death, or the last visit date serves.Estimate up to 3 years
  The duration of treatment is determined from the start date to the date of death, regardless of the cause of death. For patients still alive at the time of final analysis, the last visit date serves as both the observation endpoint and the censoring date.
Objective Response Rate（ORR） | From the start of receiving the treatment regimen in this study until the subject's disease progression and subsequent withdrawal from the study.Estimate up to 2 years
  The percentage of subjects achieving a best response of complete remission (CR) or partial remission (PR) from the start of the study treatment regimen until disease progression or withdrawal from the study, relative to the total number of subjects in the analysis set. Assessed using RECIST 1.1 criteria.
Disease Control Rate（DCR） | Estimate up to 2 years
  The proportion of subjects achieving complete remission (CR), partial remission (PR), and stable disease (SD) among all subjects.
Duration of Relief (DOR) | The time from the first assessment of tumor response as CR or PR (whichever occurs first) to the first assessment of PD or death from any cause (whichever occurs first).Estimate up to 2 years.
  The time from the first assessment of tumor response as CR or PR (whichever occurs first) to the first assessment of PD or death from any cause (whichever occurs first).
Adverse Events (AE) | about 2 years
  Incidence and grade (including serious adverse events and immunization-related adverse events), as determined by NCI-CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China